CLINICAL TRIAL: NCT02993393
Title: Faculty of Medicine Siriraj Hospital
Brief Title: A Comparative Study Between Simulation-based and Problem-based Learning in Difficult Airway Management Workshop
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mrs.Parichad Apidechakul, Nurse anesthetist, Siriraj Hospital
Other Study IDs: 369/2558(EC3)
Record Dates: First submitted 2016-12-09; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Education
Keywords: Simulation Training [I02.903.847]; Problem-Based Learning [F02.463.425.720]
MeSH Terms: interventions — Supervised Machine Learning

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Teachers: Anesthesiologists who have involved in SBL and PBL with more than 3 years of experience in teaching
  Interventions: Other: Teacher
- Students: Students were nurse anesthetist students in the academic years of 2015
  Interventions: Other: Student

INTERVENTIONS:
Other: Teacher — The teachers' questionnaire based on table of specification of the learning contents, consisted of 4 parts: airway evaluation, patient preparation, strategic planning and follow up care.
  Groups: Teachers
Other: Student — The students' questionnaire comprised 3 parts: learning content, process and evaluation.
  Groups: Students

SUMMARY:
Abstract Background and Goal of study Teaching and learning in airway management are essential in anesthetic field. Though simulation-based and problem-based learning are sophisticated learning tool, neither of them manifests the superior benefit. We would like to compare the teachers' and students' attitudes on these two learning methods.

Material and Methods After IRB approval No. 369/2558(EC3). A prospective, questionnaires-based study was performed amongst volunteered, consent-signed, 10 anesthesiologists and 40 nurse anesthetist students. After stratified randomization, ten students simultaneously attended either SBL or PBL course one at a time. Six weeks later, a crossover technique was applied for both groups. At the end of project, teachers and students had to response to Likert's scale questionnaires.

The teachers' questionnaire based on table of specification of the learning contents, consisted of 4 parts: airway evaluation, patient preparation, strategic planning and follow up care. The students' questionnaire comprised 3 parts: learning content, process and evaluation.

The validation of the questionnaire was determined by three board-certified anesthesiologists. The index of item objective congruence was 0.80 and 0.82 with Cronbach's Alpha of 0.97 and 0.92 respectively.

DETAILED DESCRIPTION:
Introduction Currently, teachers have emphasized the instructional strategies and enthusiasm in critical thinking to students to understand the educational course1. As coaching mentors, they search for innovative teaching models to reach the learning target 2. In anesthesia, a training program of nurse students involves several teaching methods such as seminars, journal clubs as well as topic, didactic, simulation and problem-based learning 13, 14.

Simulation-based learning in medicine utilizes aides such as manikins or actors to replicate clinical scenarios. It yields the acquisition of skills through deliberate practice rather than an apprentice style of learning 22. However, problem-based learning is a small group discussions where students are active, learner-centered, or self-directed learning to the topic assignments. Teachers play role as moderators or facilitators 21.

Teaching and learning in airway management are essential in anesthetic field. The personnel need to be keen both basic and advance knowledge owing to its applications to the benefits of patients' life. At present, the diversity of learning techniques (PBL and SBL) allows sophisticated devices as an interactive learning tool to cope with all difficulties in details.

Nevertheless, neither PBL nor SBL manifests the superior benefit of instructional process and learning content xx. Chin KL, et al. (2014) concluded that simulation was superior to case-based learning in teaching diabetic ketoacidosis and thyroid storm to the final-year, undergraduate pharmacy students. Randolph H, et al. (2006) revealed that students who learned critical assessment and management skills using full-scale, high- fidelity simulation, performed better than students who acquired similar skills in an interactive problem-based learning format.

As either PBL or SBL on difficult airway management is based upon the same table of specifications and experienced instructors. We would like to compare the teachers' and students' attitudes on these two learning methods.

Objectives To compare between PBL and SBL in terms of learning content, instructional and evaluation methods

Material and Methods After IRB approval No. 369/2558(EC3). A prospective, questionnaires-based study was performed amongst 40 volunteered, consent-signed nurse anesthetist students. The inclusion criteria for teachers were anesthesiologists who have involved in SBL and PBL with more than 3 years of experience in teaching. The inclusion criteria for students were nurse anesthetist students in the academic years of 2015. The exclusion criteria of both groups were ones who did not fit all qualifications.

After stratified randomization, ten nurse anesthetist students attended either SBL or PBL course one at a time. The one-day workshops were performed simultaneously. Six weeks later, a crossover technique was applied for both groups. At the end of project, teachers and students had to response to Likert's scale questionnaires: 4 = very suitable, 3 = suitable, 2 = unsuitable, 1 = very unsuitable.

The teachers' questionnaire based on table of specification of the learning contents, consisted of 4 parts: airway evaluation (history taking and physical examination), patient preparation (equipments and experienced helpers), 5 strategic planning (facemask ventilation, supraglottic airway device, laryngoscopy, tracheal intubation and failed intubation) and follow up care (documentation and informative advice).

On the other hand, the students' questionnaires comprised 3 parts: learning content, process and evaluation.

The correctness and appropriateness of the questionnaires (content validity) were determined by three board-certified anesthesiologists who had at least ten year experiences in anesthesia and were not involved in the project. The tryout was performed by ten novice nurse anesthetists and five anesthesiologists on students' and teachers' matters respectively. The index of item objective congruence was 0.80 and 0.82 with Cronbach's Alpha of 0.97 and 0.92 respectively. We used percentage, mean, standard deviation and student t-Test for data analysis at the significant level of 0.05 with 95% confident interval.

ELIGIBILITY:
Inclusion Criteria:

* anesthesiologists who have involved in SBL and PBL with more than 3 years of experience in teaching.
* nurse anesthetist students in the academic years of 2015.

Exclusion Criteria:

* ones who did not fit all qualifications.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: anesthesiologists who have involved in SBL and PBL with more than 3 years of experience in teaching.
  nurse anesthetist students
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Student's point of view | 1 year
  Likert's scale questionnaires 4 = very suitable, 3 = suitable, 2 = unsuitable, 1 = very unsuitable.

SECONDARY OUTCOMES:
Teacher's point of view | 1 year
  Likert's scale questionnaires 4 = very suitable, 3 = suitable, 2 = unsuitable, 1 = very unsuitable.

CONTACTS AND LOCATIONS:
Overall Officials: Mrs.Parichad Apidechakul, MPA. B.Ns., Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Siriraj hospital
Locations (1):
- Parichad Apidechakul, Nonthaburi, Changwat Nonthaburi, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Reilly A, Spratt C. The perceptions of undergraduate student nurses of high-fidelity simulation-based learning: a case report from the University of Tasmania. Nurse Educ Today. 2007 Aug;27(6):542-50. doi: 10.1016/j.nedt.2006.08.015. Epub 2006 Oct 25. PMID 17069935
- [Result] Rowan CJ, McCourt C, Beake S. Problem based learning in midwifery--the students' perspective. Nurse Educ Today. 2008 Jan;28(1):93-9. doi: 10.1016/j.nedt.2007.02.014. Epub 2007 May 11. PMID 17499395
- [Result] Lorello GR, Cook DA, Johnson RL, Brydges R. Simulation-based training in anaesthesiology: a systematic review and meta-analysis. Br J Anaesth. 2014 Feb;112(2):231-45. doi: 10.1093/bja/aet414. Epub 2013 Dec 23. PMID 24368556
- [Result] Chilkoti G, Mohta M, Wadhwa R, Saxena AK. Problem-based learning research in anesthesia teaching: current status and future perspective. Anesthesiol Res Pract. 2014;2014:263948. doi: 10.1155/2014/263948. Epub 2014 May 29. PMID 24982673
- [Result] Al-Elq AH. Simulation-based medical teaching and learning. J Family Community Med. 2010 Jan;17(1):35-40. doi: 10.4103/1319-1683.68787. PMID 22022669